CLINICAL TRIAL: NCT06432166
Title: 2-Hydroxybenzylamine (2-HOBA) Phase 1b/2a Proof-of Concept, Dose-Finding, Biomarker Study in Early Alzheimer's Patients
Brief Title: 2-Hydroxybenzylamine (2-HOBA) Study in Early Alzheimer's Patients
Acronym: 2-HOBA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MTI Biotech Inc (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI2024-CS01; RC-201910-2019696 (Other Grant/Funding Number: Alzheimer's Drug Discovery Foundation); IRB 231544 (Other: VUMC IRB)
Record Dates: First submitted 2024-05-14; First posted 2024-05-29 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Intervention Model Description: A phase 1b/2a, randomized, double-blind, placebo-controlled, parallel group dose finding and biomarker study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment will be supplied in capsules of the same size and color.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo treatment TID for 16 weeks.
  Interventions: Other: Placebo
- 250 mg 2-HOBA acetate (Active Comparator): 250 mg of 2-hydroxybenzylamine (2-HOBA) acetate TID for 16 weeks.
  Interventions: Drug: 2-hydroxybenzylamine acetate
- 500 mg 2-HOBA acetate (Active Comparator): 500 mg of 2-hydroxybenzylamine (2-HOBA) acetate TID for 16 weeks.
  Interventions: Drug: 2-hydroxybenzylamine acetate
- 750 mg 2-HOBA acetate (Active Comparator): 750 mg of 2-hydroxybenzylamine (2-HOBA) acetate TID for 16 weeks.
  Interventions: Drug: 2-hydroxybenzylamine acetate

INTERVENTIONS:
Drug: 2-hydroxybenzylamine acetate — 2-hydroxybenzylamine acetate (2-HOBA) is taken three times per day for 16 weeks
  Other Names: 2-HOBA
  Arms: 250 mg 2-HOBA acetate; 500 mg 2-HOBA acetate; 750 mg 2-HOBA acetate
Other: Placebo — Placebo taken three times per day for 16 weeks.
  Arms: Placebo

SUMMARY:
Investigators propose a phase 1b/2a, randomized, double-blind, placebo-controlled, parallel group dose finding and biomarker study to evaluate the safety, tolerability, and biomarker activity of 2-HOBA in 48 MCI/AD participants. Participants will be randomized 1:1:1:1 to receive 250, 500, 750 mg 2-HOBA acetate TID or placebo for 16 weeks. Blood and cerebral spinal fluid (CSF) will be collected to measure markers of protein modification by dicarbonyls (IsoLGs- & MDA), pTau-181, YKL-40, and NF-L.

DETAILED DESCRIPTION:
This is a phase 1b/2a, randomized, double-blind, placebo-controlled, parallel group dose finding and biomarker study to evaluate the safety, tolerability, and biomarker activity of 2-HOBA in 48 MCI/AD participants. Participants will be randomized 1:1:1:1 to receive 250, 500, 750 mg 2-HOBA acetate TID or placebo for 16 weeks. Blood and CSF will be collected to measure markers of protein modification by dicarbonyls (IsoLGs- & MDA), pTau-181, YKL-40, and NF-L. Investigators anticipate screening 120 subjects to randomize up to 60 subjects with the goal of 48 patients completing the study (allowing for up to 25% dropout) for the 16-week study.

The primary aims of this project are to 1) Provide proof-of-concept that 2-HOBA protects proteins from covalent modification by inhibiting lysine-reacting dicarbonyls in the human brain. Investigators hypothesize that 16 weeks of 2-HOBA treatment will significantly reduce CSF levels of the dilysyl-MDA and IsoLG adduct of CSF proteins in a dose-responsive relationship. 2) Evaluate whether 2-HOBA is safe for extended use in patients with early AD. Investigators hypothesize that 2-HOBA will be safe and well tolerated through 16 weeks of use. Tolerability will be assessed by monitoring symptoms, adverse events, vital signs, ECG, and safety labs during the study.

The secondary aims are to evaluate the effect of 2-HOBA treatment on AD biomarkers, brain inflammation, disease severity, and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

MCI due to AD:

1. Male or female, aged 55-85 years (both inclusive) at the time of signing informed consent.
2. Participant must have a subjective memory concern as reported by participant, study partner, or clinician.
3. Mini-Mental State Exam31 score between 24 and 30, inclusive
4. Clinical Dementia Rating (CDR)32 Global = 0.5. Memory Box score must be at least 0.5.

Mild AD:

1. Male or female, aged 55-85 years (both inclusive) at the time of signing informed consent.
2. Mild dementia of the Alzheimer's type according to the NIA-AA 2018 criteria.
3. CDR global score of 0.5 and CDR of 0.5 or more in at least one of the three instrumental activities of daily living categories (personal care, home & hobbies, community affairs) Or CDR global score of 1.0
4. MMSE ≥20

Additional Inclusion Criteria for Both Diagnoses:

1. Age 55-85 (inclusive)
2. Abnormal memory function documented by scoring within the education adjusted ranges on the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised:

   * Less than or equal to 11 for 16 or more years of education
   * Less than or equal to 9 for 8 - 15 years of education
   * Less than or equal to 6 for 0 - 7 years of education
3. Amyloid positivity established using the C2N Precivity2 Plasma test (Aβ42/40 plus p- tau217/np-tau217. (This test uses a statistical algorithm to integrate a patient's Aβ42/40 Ratio and p-Tau217 Ratio to calculate the Amyloid Probability Score 2 (APS2) and determines whether a patient is positive or negative for brain amyloid deposition based on a binary cutoff value).
4. Stable permitted medications for 4 weeks or longer as specified in Section 4.6.3, including:

   a. Memantine and cholinesterase inhibitors are allowable if stable for 12 weeks prior to screen.
5. Geriatric Depression Scale33 score of less than or equal to 14.
6. Study Partner is available who has frequent contact with the participant (e.g., an average of 10 hours per week or more) and can accompany the participant to most visits to answer questions about the participant.
7. Adequate visual and auditory acuity to allow neuropsychological testing.
8. Good general health with no additional diseases/disorders expected to interfere with the study.
9. Participant is not pregnant, lactating, or of childbearing potential (i.e., women must be two years post-menopausal or surgically sterile).
10. Completed six grades of education or has a good work history.
11. Must speak English fluently.
12. Provide written informed consent. Participants must have the capacity to consent.

Exclusion Criteria:

1. Any other significant neurologic disease including Parkinson's disease, multi- infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
2. Major depression, bipolar disorder as described in DSM-V within the past 1 year or psychotic features, agitation, or behavioral problems within 3 months, which could lead to difficulty complying with the protocol.
3. History of schizophrenia (DSM V criteria).
4. History of alcohol or substance abuse or dependence within the past 2 years (DSM V criteria).
5. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic (Class C defined by Child-Pugh criteria), endocrine, or other systemic disease in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results, or the participant's ability to participate in the study.
6. Has had a history within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment.
7. Clinically significant abnormalities in B12 or TFTs that might interfere with the study. A low B12 is exclusionary, unless the required follow-up labs (homocysteine (HC) and methylmalonic acid (MMA) indicate that it is not physiologically significant.
8. Clinically significant abnormalities in screening laboratories or ECG.
9. Residence in a skilled nursing facility.
10. Use of any excluded medication as described in Section 6.10, including:

    * Use centrally acting anti-cholinergic drugs.
    * Use of any investigational drugs within 4 weeks or 5 half-lives, whichever is longer, prior to screening.
11. A current blood clotting or bleeding disorder, or significantly abnormal PT or PTT at screening.
12. Contraindications for MRI studies, including claustrophobia, the presence of metal(ferromagnetic) implants, or cardiac pacemaker.
13. Participants whom the Site PI deems to be otherwise ineligible.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability (adverse events) | Baseline to week 16
  Rates of adverse events will be compared between active and placebo arms and presented as summary statistics.
Change in dicarbonyl protein adducts | Baseline to week 16
  Change in CSF levels of the dilysyl-malondialdehyde crosslink and the lysyl-levuglandin adduct of CSF proteins in a dose-responsive relationship

SECONDARY OUTCOMES:
Compliance | Baseline to week 16
  Treatment compliance will be assessed through pill counts at Week 8 and 16
Measurement of biomarker, p-Tau181 | Baseline to week 16
  Change in phosphorylated-Tau-181 levels in CSF and plasma:
Measurement biomarker, human cartilage glycoprotein 39 (YKL-4) | Baseline to week 16
  Change in plasma concentration of human cartilage glycoprotein 39 (YKL-4)
Measurment of biomarker, neurofilaments light chain protein (NF-L) | Baseline to week 16
  Change in the concentration of neurofilaments light chain protein (NF-L) in CSF and plasma
Measurement of biomarker, F2-Isoprostanes | Baseline to week 16
  Change in concentration F2-Isoprostanes in plasma and urine:
Measurement of biomarker, 8-hydroxy-2'-deoxyguanosine | Baseline to week 16
  Change in concentration of 8-hydroxy-2'-deoxyguanosine in plasma

OTHER OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline to Week 16
  Change in the total score for the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Activities of Daily Living (ADL) | Baseline to Week 16
  For Activities of Daily Living (ADLs), the Alzheimer's disease Cooperative Study Activities of Daily Living (ADCS-ADL) scale to assess the competence of participants in basic and instrumental ADLs will be utilized. A lower score indicates greater functional impairment.
Quantitative Electroencephalography (EEG) | Baseline to Week 16
  The change participants' electrical brain activity will be monitored using noninvasive scalp electrodes. Event-related potentials (ERP), or time-locked EEG, will be used to evaluate cognitive processes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newhouse, M.D., Principal Investigator — Vanderbilt University Medical Center; John A. Rathmacher, Ph.D., Principal Investigator — MTI Biotech Inc
Locations (1):
- Center for Cognitive Medicine, Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No